CLINICAL TRIAL: NCT01295151
Title: Randomised-controlled Trial of Switching to Alternative Tumour-necrosis Factor (TNF)-Blocking Drugs or Abatacept or Rituximab in Patients With Rheumatoid Arthritis Who Have Failed an Initial TNF-blocking Drug
Brief Title: SWITCH Clinical Trial for Patients With Rheumatoid Arthritis Who Have Failed an Initial TNF-blocking Drug.
Acronym: SWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Julia Brown (Other)
Responsible Party: Sponsor-Investigator, Julia Brown, Director of Leeds Institute of Clinical Trials Research, University of Leeds
Organization: University of Leeds (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RR10/9589; 2010-023880-17 (EudraCT Number)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Abatacept; Rituximab; Adalimumab; Certolizumab Pegol; Infliximab; golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TNF-blocking drug (Experimental)
  Interventions: Drug: Etanercept; Drug: Adalimumab; Drug: Certolizumab Pegol; Drug: Infliximab; Drug: Golimumab
- Abatacept (Experimental)
  Interventions: Drug: Abatacept
- Rituximab (Active Comparator)
  Interventions: Biological: Rituximab

INTERVENTIONS:
Drug: Etanercept — Etanercept will be administered at a dose of 50mg by subcutaneous injection per week for a total of 12 weeks. Further treatment will be prescribed at the discretion of the treating clinician.
  The patient will be taught how to administer the subcutaneous injection and injections will be monitored by the hospital until the patient is proficient with the technique.
  Arms: TNF-blocking drug
Drug: Abatacept — Abatacept will be administered at a dose determined by body weight:
  Body Weight (kg) Dose (mg) < 60kg = 500 mg
  > or equal to 60kg and < or equal to 100kg = 750 mg > 100 kg = 1000mg
  The intravenous infusions will be administered in clinic on days 1, 15, 29 and every 28 days thereafter for a minimum of 24 weeks. Further treatment will be prescribed at the discretion of the treating clinician.
  Arms: Abatacept
Biological: Rituximab — Rituximab will be given at a dose of 1000mg; 2 intravenous infusions will be administered at days 0 (week 0) and 15 (week 2).
  In line with standard practice, a patient who loses an initial response with a DAS28 increase of at least 0.6 may receive a further cycle of rituximab at the discretion of the treating clinician.
  Prior to receiving rituximab, intravenous methylprednisolone 100mg will also be given.
  Arms: Rituximab
Drug: Adalimumab — Adalimumab will be given at a dose of 40mg by subcutaneous injection every two weeks for a minimum of 12 weeks. Further treatment will be prescribed at the discretion of the treating clinician.
  The patient will be taught how to administer the subcutaneous injection and injections will be monitored by the hospital until the patient is proficient with the technique.
  Arms: TNF-blocking drug
Drug: Certolizumab Pegol — Certolizumab Pegol will be given at a dose of 400mg by subcutaneous injection at weeks 0, 2, 4and then at a dose of 200mg every two weeks thereafter for a minimum of 12 weeks. Further treatment will be prescribed at the discretion of the treating clinician.
  The patient will be taught how to administer the subcutaneous injection and injections will be monitored by the hospital until the patient is proficient with the technique.
  Arms: TNF-blocking drug
Drug: Infliximab — Infliximab will be given at a dose of 3mg/kg per intravenous infusion in clinic.
  The intravenous infusions will be administered at week 0, 2, 6 and then 8-weekly thereafter for a minimum of 12 weeks.
  Further treatment will be prescribed at the discretion of the treating clinician.
  Arms: TNF-blocking drug
Drug: Golimumab — Golimumab will be given at a dose of 50mg by subcutaneous injection every 4 weeks for a minimum of 24 weeks.
  Further treatment will be prescribed in line with the study protocol and following week 48, at the discretion of the treating clinician.
  The participant will be taught how to administer the subcutaneous injection and injections will be monitored according to local arrangements until the participant is proficient with the technique according to local practice.
  Arms: TNF-blocking drug

SUMMARY:
The principal aim of this study is to fill a clear knowledge gap and provide guidance for rheumatologists and reassurance to the patient group on a management challenge faced daily in rheumatology practice. Specifically, it aims to provide robust evidence on the optimal management of patients with established RA that have failed an anti-TNF therapy (the first of the biological therapies to be introduced); in particular, the investigators wish to address whether the currently licensed but non NICE-approved treatment options, TNF-blocking drug or abatacept, are equivalent to the NICE-approved treatment, rituximab. If so, the intention is to broaden treatment options and target these specific therapies to disease sub-groups.

ELIGIBILITY:
Inclusion Criteria

1. Male and female subjects aged ≥18 years at the time of signing the Informed Consent Form.
2. Patients with a diagnosis of rheumatoid arthritis as per the ACR/EULAR 2010 classification criteria (Appendix 7) confirmed at least 24 weeks prior to the screening visit.
3. Patients who have failed conventional DMARD therapy as per NICE/BSR Guidelines (49) i.e. failure of at least 2 DMARDS including MTX.
4. Patients with persistent RA disease activity despite having been treated with a current initial TNFi agent for at least 12 weeks. Active RA defined as*:

   1. Primary non-response: failing to improve DAS28 by > 1.2 (Appendix 6) or failing to achieve DAS28 ≤ 3.2 within the first 12 to 24 weeks of starting the initial TNFi.

      • This may include patients that have shown a reduction in DAS28 of > 1.2 but still demonstrate unacceptably high disease activity in the physician's judgement with evidence of an overall DAS28 of ≥ 3.2 OR
   2. Secondary non-response: defined as inefficacy to first TNFi (having demonstrated prior satisfactory response) as per clinician judgement; with intolerance not the reason for cessation of first TNFi.
5. MTX dose stable for 4 weeks prior to the screening visit and to be continued for the duration of the study.
6. Patients on NSAIDs and / or corticosteroids (oral prednisolone not exceeding 10mg daily) who have been on an unchanged regimen for at least 4 weeks prior to the screening visit and are expected to remain on a stable dose until the baseline assessments have been completed.
7. Provided written informed consent prior to any trial-specific procedures.

Exclusion Criteria

1. Major surgery (including joint surgery) within 8 weeks prior to the screening visit or planned major surgery within 52 weeks following randomization.
2. Patients with inflammatory joint disease of different origin, mixed connective tissue disease, Reiter's syndrome, psoriatic arthritis, systemic lupus erythematosus, or any arthritis with onset prior to 16 years of age.
3. Patients receiving doses of prednisolone > 10mg/day within the 4 weeks prior to the screening visit.
4. Patients receiving intra-articular or intra-muscular steroid injections within 4 weeks prior to the screening visit.
5. Patients who have previously received more than 1 TNFi drug OR any other biological therapy for the treatment of RA.
6. Patients unable or unwilling to stop treatment with a prohibited DMARD (i.e synthetic DMARD aside from MTX e.g. oral or injectable gold, chloroquine, hydroxychloroquine, cyclosporine, azathioprine, leflunomide, sulphasalazine) prior to the start of protocol treatment.
7. Treatment with any investigational drug in the last 12 weeks prior the start of protocol treatment.
8. Patients with other co-morbidity including acute, severe infections, uncontrolled diabetes, uncontrolled hypertension, unstable ischaemic heart disease, moderate/severe heart failure (Class III/IV of the New York Heart Association (NYHA) functional classification system (79)), active bowel disease, active peptic ulcer disease, recent stroke (within 12 weeks before the screening visit), or any other condition which, in the opinion of the investigator, would put the patient at risk to participate in the study or would make implementation of the protocol difficult.
9. Patients with any major episode of infection requiring hospitalisation or treatment with IV antibiotics within 12 weeks of start of treatment protocol or oral antibiotics within 4 weeks of start of protocol treatment.
10. Patients at significant risk of infection, which in the opinion of the investigator would put the patient at risk to participate in the study (e.g. leg ulceration, indwelling urinary catheter, septic joint within 52 weeks (or ever if prosthetic joint still in situ)).
11. Patients with known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections including herpes zoster (for tuberculosis and Hepatitis B and C see below), but excluding fungal infections of nail beds as per clinical judgment.
12. Patients with untreated active current or latent tuberculosis (TB). Patients should have been screened for latent TB (as per BSR guidelines) within 24 weeks prior to the screening visit and, if positive, treated following local practice guidelines prior to the start of protocol treatment.
13. Patients with active current hepatitis B and/or C infection. Patients should have been screened for hepatitis B and C within 24 weeks prior to the screening visit and if positive, excluded from the study.
14. Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.
15. Pregnancy, lactation or women of child-bearing potential (WCBP) unwilling to use an effective birth control measure (Appendix 2) whilst receiving treatment and after the last dose of protocol treatment as indicated in the relevant SmPC/IB.
16. Men whose partners are of child-bearing potential but who are unwilling to use an effective birth control measure (Appendix 2) whilst receiving treatment and after the last dose of protocol treatment as indicated in the relevant SmPC/IB.
17. Patients with known significantly impaired bone marrow function as for example significant anaemia, leukopaenia, neutropaenia or thrombocytopaenia as shown by the following laboratory values at the time of the screening visit:

    * Haemoglobin < 8.5 g/dl
    * Platelet count < 100 x 109 / L
    * White blood cell count < 2.0 x 109 / L
    * Neutrophil count < 1 x 109 / L
18. Patients with known severe hypoproteinaemia at the time of the screening visit, e.g. in nephrotic syndrome or impaired renal function, as shown by:

    * Serum Creatinine > 150 umol / L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in disease activity. | 6 months
  Change in Disease Activity Score 28 (DAS28) at 6 months (24 weeks).

SECONDARY OUTCOMES:
Reduction in disease activity. | Baseline and weeks 12, 24, 36 & 48.
  Proportion of participants who achieve a reduction in DAS28 score of greater than 1.2 from baseline at weeks 12, 24, 36 and 48 with no toxicity.
EULAR & ACR Response Scores | Baseline and weeks 12, 24, 36, 48
  EULAR Response Scores and American College of Rheumatology (ACR) Response Scores (evaluated at weeks 12, 24, 36, 48).
CDAI (Clinical disease activity index) | Baseline and weeks 12, 24, 36 & 48.
  Change in CDAI score from baseline at weeks 12, 24, 36 and 48. Proportion of participants in each CDAI category at weeks 12, 24, 36 & 48.
SDAI (Simplified Disease Activity Index) | Baseline and weeks 12, 24, 36 & 48.
  Change in SDAI score from baseline at weeks 12, 24, 36 & 48. Proportion of participants in each SDAI category at weeks 12, 24, 36 & 48.
ACR/EULAR Boolean remission rates | Baseline and weeks 12, 24, 36 & 48.
  Proportion of participants that achieve Boolean remission rate at weeks 12, 24, 36 & 48.
Quality of Life Assessments | Baseline & weeks 12, 24, 36 & 48.
  RA Quality of Life (RAQoL) score Health Assessment Questionnaire Disability Index (HAQ-DI) (also evaluated at weeks 60, 72, 84 & 96) Hospital Anxiety and Depression Scale (HADS)
Safety & Toxicity | Baseline and weeks 12, 24, 36 & 48.
  Toxicity Adverse Events & Reactions
Economic Evaluation | Baseline & weeks 12, 24, 36 & 48
  EuroQol 5-dimensions (EQ-5D) (also evaluated at weeks 60, 72, 84 & 96) Health Utilities Index (also evaluated at weeks 60, 72, 84 & 96) Health and Social Care Use & Expenditure due to Rheumatoid Arthritis (evaluated at weeks 12, 24, 36 & 48) Incremental Cost Effectiveness
Imaging (at the discretion of individual sites) | Baseline and week 48.
  Change in plain x-ray score of hands and feet (Modified Genant score - evaluated at baseline and week 48) Bone densitometry scan scores (T-scores unilateral neck of femur and lumbar spine - evaluated at baseline and week 48)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Buch, Principal Investigator — University of Leeds
Locations (1):
- Institute of Rheumatic & Musculoskeletal Medicine, Chapel Allerton Hospital, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Plein S, Erhayiem B, Fent G, Horton S, Dumitru RB, Andrews J, Greenwood JP, Emery P, Hensor EM, Baxter P, Pavitt S, Buch MH. Cardiovascular effects of biological versus conventional synthetic disease-modifying antirheumatic drug therapy in treatment-naive, early rheumatoid arthritis. Ann Rheum Dis. 2020 Nov;79(11):1414-1422. doi: 10.1136/annrheumdis-2020-217653. Epub 2020 Aug 28. PMID 32859608
- [Derived] Brown S, Everett CC, Naraghi K, Davies C, Dawkins B, Hulme C, McCabe C, Pavitt S, Emery P, Sharples L, Buch MH. Alternative tumour necrosis factor inhibitors (TNFi) or abatacept or rituximab following failure of initial TNFi in rheumatoid arthritis: the SWITCH RCT. Health Technol Assess. 2018 Jun;22(34):1-280. doi: 10.3310/hta22340. PMID 29900829
- [Derived] Navarro Coy NC, Brown S, Bosworth A, Davies CT, Emery P, Everett CC, Fernandez C, Gray JC, Hartley S, Hulme C, Keenan AM, McCabe C, Redmond A, Reynolds C, Scott D, Sharples LD, Pavitt S, Buch MH. The 'Switch' study protocol: a randomised-controlled trial of switching to an alternative tumour-necrosis factor (TNF)-inhibitor drug or abatacept or rituximab in patients with rheumatoid arthritis who have failed an initial TNF-inhibitor drug. BMC Musculoskelet Disord. 2014 Dec 23;15:452. doi: 10.1186/1471-2474-15-452. PMID 25539805